CLINICAL TRIAL: NCT07398417
Title: A Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Assess the Efficacy and Safety of AXS-14 in the Management of Fibromyalgia
Brief Title: Fibromyalgia Response With Esreboxetine Evaluated Using a Randomized Withdrawal Research Design
Acronym: FORWARD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-14-FM-301
Record Dates: First submitted 2026-02-04; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Central Sensitization; Allodynia; Hyperalgesia; Hypersensitivity to sensory stimuli; Inhibitor of the norepinephrine transporter (NET); Esreboxetine; AXS-14; Axsome; Norepinephrine reuptake inhibitor
MeSH Terms: conditions — Fibromyalgia; Hyperalgesia | interventions — esreboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-14 (esreboxetine) (Experimental): * Up to 12 weeks in the open-label period;
  * Up to 12 weeks in the randomized double-blind period (if applicable)
  Interventions: Drug: AXS-14 (Esreboxetine)
- Placebo (Placebo Comparator): • Up to 12 weeks in the randomized double-blind period (if applicable)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-14 (Esreboxetine) — AXS-14 tablets taken once daily
  Arms: AXS-14 (esreboxetine)
Drug: Placebo — Placebo tablets taken once daily
  Arms: Placebo

SUMMARY:
The study is a Phase 3, double-blind, placebo-controlled, randomized withdrawal study to assess the efficacy and safety of AXS-14 in the management of fibromyalgia.

DETAILED DESCRIPTION:
This study is a multi-center trial consisting of a 12-week open-label treatment period (OLP), followed by a 12-week double-blind, placebo-controlled, randomized withdrawal period (DBRWP). During the OLP, subjects receive open-label AXS-14. Subjects achieving treatment response will be randomized into the DBRWP in a 1:1 ratio to either continue on AXS-14 or switch to placebo for up to 12 weeks or until a loss of therapeutic response occurs.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of fibromyalgia based on the 2016 ACR diagnostic criteria.
* Male or female, ≥18 years of age.
* Provides written informed consent to participate in the study before conducting any study procedures.

Exclusion Criteria:

* Previous participation in a clinical trial with reboxetine or esreboxetine or currently receiving treatment with reboxetine for any condition.
* Unable to comply with study procedures.
* Medically inappropriate for study participation in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to loss of therapeutic response | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Cromwell, Connecticut
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Overland Park, Kansas
  - Clinical Research Site, Louisville, Kentucky
  - Clinical Research Site, Prairieville, Louisiana
  - Clinical Research Site, Springfield, Missouri
  - Clinical Research Site, Town and Country, Missouri
  - Clinical Research Site, Tulsa, Oklahoma
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Prosper, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com